CLINICAL TRIAL: NCT06171490
Title: A Multi-center, Randomized, Controlled, Partially Blinded Study to Assess the Pharmacokinetics and Comparative Bioavailability of Nicotine From Two Variants of Nicotine Pouch 2.0 (NP2), 4mg and 6mg, Compared to Nicotine Lozenge 4mg and Nicotine Gum 4mg in Adult Cigarette Smokers
Brief Title: Pharmacokinetics and Comparative Bioavailability of Nicotine From Two Variants of NP2, NP2-4mg and NP2-6mg, Compared to Nicotine Lozenge 4mg (Loz-4mg) and Nicotine Gum 4mg (Gum-4mg)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PZ-PK-03-CAN
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Tobacco Use
Keywords: Nicotine; Nicotine-containing products; Tobacco; Pharmacokinetics
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: The study will be conducted with 4 periods and 4 sequences in a Williams design (crossover).
Who Masked: Participant, Investigator
Masking Description: This is a partially blinded study. The Investigator and subjects will be blinded to the randomized sequence and to the variants of the investigational product (IP). In contrast, the pharmacy staff will not be blinded to the randomized sequence and to the variants of the IP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Product Sequence 1 (Active Comparator): From Day 1 to Day 4, after at least 23 hours of abstinence from any nicotine/tobacco containing products, subjects will use one of the four investigational products according to randomized product use sequence and as instructed by the investigational site personnel.
  The list of possible sequences are:
  NP2-4mg; NP2-6mg; Loz-4mg; Gum-4mg / NP2-6mg; Gum-4mg; NP2-4mg; Loz-4mg / Gum-4mg; Loz-4mg; NP2-6mg; NP2-4mg / Loz-4mg; NP2-4mg; Gum-4mg; NP2-6mg
  Interventions: Other: NP2-4mg; Other: NP2-6 mg; Other: Loz-4mg; Other: Gum-4mg
- Product Sequence 2 (Active Comparator): From Day 1 to Day 4, after at least 23 hours of abstinence from any nicotine/tobacco containing products, subjects will use one of the four investigational products according to randomized product use sequence and as instructed by the investigational site personnel.
  The list of possible sequences are:
  NP2-4mg; NP2-6mg; Loz-4mg; Gum-4mg / NP2-6mg; Gum-4mg; NP2-4mg; Loz-4mg / Gum-4mg; Loz-4mg; NP2-6mg; NP2-4mg / Loz-4mg; NP2-4mg; Gum-4mg; NP2-6mg
  Interventions: Other: NP2-4mg; Other: NP2-6 mg; Other: Loz-4mg; Other: Gum-4mg
- Product Sequence 3 (Active Comparator): From Day 1 to Day 4, after at least 23 hours of abstinence from any nicotine/tobacco containing products, subjects will use one of the four investigational products according to randomized product use sequence and as instructed by the investigational site personnel.
  The list of possible sequences are:
  NP2-4mg; NP2-6mg; Loz-4mg; Gum-4mg / NP2-6mg; Gum-4mg; NP2-4mg; Loz-4mg / Gum-4mg; Loz-4mg; NP2-6mg; NP2-4mg / Loz-4mg; NP2-4mg; Gum-4mg; NP2-6mg
  Interventions: Other: NP2-4mg; Other: NP2-6 mg; Other: Loz-4mg; Other: Gum-4mg
- Product Sequence 4 (Active Comparator): From Day 1 to Day 4, after at least 23 hours of abstinence from any nicotine/tobacco containing products, subjects will use one of the four investigational products according to randomized product use sequence and as instructed by the investigational site personnel.
  The list of possible sequences are:
  NP2-4mg; NP2-6mg; Loz-4mg; Gum-4mg / NP2-6mg; Gum-4mg; NP2-4mg; Loz-4mg / Gum-4mg; Loz-4mg; NP2-6mg; NP2-4mg / Loz-4mg; NP2-4mg; Gum-4mg; NP2-6mg
  Interventions: Other: NP2-4mg; Other: NP2-6 mg; Other: Loz-4mg; Other: Gum-4mg

INTERVENTIONS:
Other: NP2-4mg — NP2-4 mg is a new product containing tobacco-derived nicotine.
Other: NP2-6 mg — NP2-6 mg is a new product containing tobacco-derived nicotine.
Other: Loz-4mg — The Loz-4mg reference product is a commercially available 4mg nicotine lozenge.
Other: Gum-4mg — The Gum-4mg reference product is a commercially available 4mg nicotine gum.

SUMMARY:
This is a multi-center, randomized, controlled, partially blinded study to assess the pharmacokinetics and comparative bioavailability of nicotine from two variants of NP2 (4 and 6 mg) in comparison with Loz-4mg and Gum-4mg in adult cigarette smokers. The subjects will be blinded to the randomized sequence and will be blinded to the variants of NP2 they will receive. The study will be conducted with 4 periods and 4 sequences in a Williams design (crossover).

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed the ICF and is able to understand the information provided in the ICF.
* Subject has smoked on a daily basis for at least the last 18 months prior to the Screening visit.
* Subject has smoked on average ≥10 commercially available regular CIG/day over the last 4 weeks. Smoking status will be verified based on a urinary cotinine test (cotinine ≥200 ng/mL).
* Subject is healthy as judged by the Investigator based on available assessments from the screening period (e.g., safety laboratory, spirometry, vital signs, physical examination, ECG, and medical history).

Exclusion Criteria:

* Subject has reasons other than medical (e.g., psychological, social reason) not to be part of the study, as determined by the Investigator.
* Subject is legally incompetent, or physically or mentally incapable of giving consent (e.g., emergency situation, under guardianship, prisoners).
* Subject has a clinically relevant disease which requires medication or any other medical condition including abnormal spirometry, safety laboratory, as determined by the Investigator.
* Subject presents difficulty with venipuncture and/or poor venous access.
* Subject has an oromucosal or dental condition, which may affect the use of the investigational products, as determined by the Investigator or subject has orthodontic braces and retention wire (could likely interfere with the gum dosing).
* Subject has medical conditions which require, or will require during the study, a medical intervention (e.g., start of treatment, surgery, hospitalization).
* Presence of fever (body temperature >37.5°C) (e.g., a fever associated with a symptomatic viral or bacterial infection) within 2 weeks prior to dosing.
* Subject has a Hemoglobin level < 11.0 g/dL for females and < 12.0 g/dL for males at the Screening.
* Subject uses medication or any substance that aids in smoking cessation.
* Subject postponed the decision to quit using tobaccoor nicotine-containing products in order to participate in this study.
* Subject previously attempted to quit using tobacco- or nicotine-containing products within 28 days prior to the first study product administration.
* Subject has donated plasma within seven days prior to Screening or has donated or lost 450 mL or more of whole blood within 8 weeks prior to Screening for males, and in the 12 weeks prior to Screening for females.
* Subject has a known sensitivity or allergy to any of the investigational products, or ingredients.
* Subject has a positive serology test for HIV 1/2, Hepatitis B, Hepatitis C.
* Subject has a history of alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
* Subject has a positive urine drug test. Investigator will assess whether THC positive subjects are eligible for participation in the study.
* Subject has a positive alcohol breath test.
* Subject or one of their family members is a current or former employee of the tobacco industry.
* Subject or one of their family members a is an employee of the investigational site or of any other parties involved in the study.
* Subject has participated in another clinical study within 30 days prior to the Screening Visit or concomitantly participates in an investigational study involving no drug or device administration.
* Subject has been previously screened or enrolled in this study (except alternate subjects).
* For women only: subject is pregnant (does not have negative pregnancy tests at Screening Visit and at Admission) or is a lactating female.
* For women of childbearing potential only: subject does not agree to use an acceptable method of effective contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Measured from start of product use to 24 hours
  To measure Cmax following use of the investigational products and reference products
Area under the observed concentration-time curve (AUC) from start of product use (T0) to timepoint of last quantifiable concentration [AUC0-last] and extrapolated to infinity [AUC0-infinity] | Measured from start of product use (T0) to 2 minutes, to 4 minutes, to 10 hours, to time of last quantifiable concentration.
  To measure the area under the background-corrected concentration-time curve (AUC) from start of product use
Ratio of [AUC0-last] and [AUC0-infinity] | Measured from start of product use to 24 hours
  To measure the ratio of [AUC0-last] and [AUC0-infinity]
Time to the observed maximum concentration [Tmax] | Measured from start of product use to 24 hours
  To measure the maximum ratio of background-corrected concentration over time, from T0 (excluded) to Tmax (included)
Elimination rate constant [kel] | Measured from start of product use to 24 hours
  To measure the fraction of nicotine eliminated per unit of time, following use of the investigational products and reference products
Half-life of nicotine [t1/2] | Measured from start of product use to 24 hours
  To measure the half-life of nicotine, following use of the investigational products and reference products

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.
Locations (2):
- Canada (2):
  - Pharma Medica Research Inc., Toronto, Ontario
  - Syneos Health Clinique Inc., Québec